CLINICAL TRIAL: NCT05717959
Title: Efficacy of Oropharyngeal Exercises for Patients With Obstructive Sleep Apnea Using Mandibular Advancement Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-ER-111-222
Record Dates: First submitted 2022-12-01; First posted 2023-02-08 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: Obstructive Sleep Apnea; Mandibular advancement device; oropharyngeal exercises
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): We conducted a once a week, 12-week-intervention of Oropharyngeal Exercises and Mandibular advancement device
  Interventions: Behavioral: Oropharyngeal Exercises
- control group (Sham Comparator): Mandibular advancement device
  Interventions: Behavioral: Oropharyngeal Exercises

INTERVENTIONS:
Behavioral: Oropharyngeal Exercises — Oropharyngeal Exercises

SUMMARY:
Combined treatment with MAD and OE for adult patients with obstructive sleep apnea can significantly (i) improve muscle strength and endurance; (ii) reduce the severity of sleep apnea.

DETAILED DESCRIPTION:
Background: Obstructive Sleep Apnea (OSA) is a sleeping disorder with recurrent upper airway obstruction during sleep. Patients with OSA often suffer from daytime sleepiness, snoring, and interrupted breathing during sleep. The etiology of OSA can divide into anatomical causes, including narrow, crowded, or easily collapsible upper airway, and non-anatomical causes, including low respiratory arousal threshold, ineffective or reduced pharyngeal dilator muscle activity during sleep, and unstable ventilatory control. A mandibular advancement device (MAD) is one of the treatment options for mild to moderate OSA patients. Oropharyngeal exercises (OE) are a novel intervention targeted at internal/external tongue muscle training with significant improvements in the muscle tension and severity of OSA. The efficacy of combined treatment with MAD and OE has not been investigated. Thus, the present study aims to determine the effectiveness of combing MAD and OE by assessing the tongue function and severity of OSA in patients with OSA.

Methods: A total of 20 participants using MAD for OSA were included in the study. Participants will be divided into two groups: the treatment group with the 12-week OE. OE consists of one to three times 30-minute sessions per day, 3 to 5 days per week for 12 weeks. The weekly clinic visits are required to adjust the intensity of the home exercise program and monitor the training progress. The participants in two groups will receive polysomnography (PSG) test, tongue muscle strength, and endurance testing, at baseline and after the intervention.

Expected results: Combined treatment with MAD and OE for adult patients with mild to moderate obstructive sleep apnea can significantly (i) improve muscle strength and endurance; (ii) reduce the severity of sleep apnea

ELIGIBILITY:
Inclusion Criteria:

* OSA patients
* aged over 20 years old
* wearing a MAD

Exclusion Criteria:

* Body Mass Index (BMI) ≧ 35
* Pregnancy
* Severe obstructive or restrictive lung disease
* Exercise with high-risk cardiovascular disease
* History of central or peripheral neurological disease resulting in an inability to perform exercise prescriptions
* Musculoskeletal or psychological disorders that prevent the performance of exercise prescriptions
* Chronic illnesses that are ongoing or not yet controlled

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea -index | Baseline to 12 weeks
  Assessed using Polysomnography (PSG). The average apnea and hypopnea events per hour, oxygen saturation index and the snoring index will be obtained during the sleep test(PSG)

SECONDARY OUTCOMES:
Tongue muscle strength | Baseline to 12 weeks
  The maximal muscle strength of genioglossus muscles using The Iowa Oral Performance Instrument (IOPI) system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA) (kPa)
Tongue muscle endurance | Baseline to 12 weeks
  The endurance of the genioglossus muscles using The Iowa Oral Performance Instrument (IOPI) system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA) (in seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Ching Hsia Hung, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No